CLINICAL TRIAL: NCT02356016
Title: Effects of Whole-body Electromyostimulation and Dietary Supplements on "Sarcopenic Obesity" in Elderly Females Living in the Community
Brief Title: Effects of Whole-body Electromyostimulation and Dietary Supplements on "Sarcopenic Obesity"
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: University of Erlangen-Nürnberg (Other); Bavarian Research Foundation, Munich, Germany (Unknown); miha bodytec, Gersthofen, Germany (Unknown); Physiomed, Laipersdorf, Germany (Unknown); Siemens AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FORMOsA P2 TP3
Record Dates: First submitted 2015-01-21; First posted 2015-02-05 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Sarcopenic Obesity
Keywords: Sarcopenic Obesity; community dwelling elderly women; electromyostimulation; exercise; dietary supplements
MeSH Terms: conditions — Motor Activity | interventions — Dietary Supplements; Nutrition Assessment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whole body Electromyostimulation (WB-EMS) (Active Comparator): 18 min of WB-EMS/week (one session/week)
  Interventions: Behavioral: WB-EMS Intervention
- WB-EMS and Nutritional Supplements (Active Comparator): 18 min of WB-EMS/week (one session/week) and supplements with high protein (Leucin) contents
  Interventions: Behavioral: WB-EMS-Intervention and dietary supplementation
- Control (Sham Comparator): Monthly dietary counseling for 6 months
  Interventions: Other: control (dietary counseling)

INTERVENTIONS:
Behavioral: WB-EMS Intervention — Supervised WB-EMS Intervention 18 min/session (one session/week) and monthly dietary counseling for 6 months
  Arms: Whole body Electromyostimulation (WB-EMS)
Behavioral: WB-EMS-Intervention and dietary supplementation — Supervised WB-EMS Intervention and dietary supplementation and monthly dietary counseling for 6 months
  Arms: WB-EMS and Nutritional Supplements
Other: control (dietary counseling) — Monthly dietary counseling only
  Arms: Control

SUMMARY:
The aim of the study is to determine the effect of whole body electromyostimulation (WB-EMS) and/or nutritional on body composition and functional tasks in elderly females with sarcopenic obesity. Seventy-five, non-sportive, independently living women 70 years and older with Sarcopenic Obesity were randomly assigned to either a WB-EMS group ( n=25), a WB-EMS/nutritional supplements (n=25) or a semi-active control group (an=25). The WB-EMS protocol applied one session of 18 min/week of WB-EMS (bipolar, 85 Hz). Nutritional strategy based on a high protein supplement.

ELIGIBILITY:
Inclusion Criteria:

* community dwelling
* Sarcopenic Obesity

Exclusion Criteria:

* exercising more than 60 min/week
* more than 4 weeks absent during the interventional period,
* injuries (i.e. hip TotalEndoProsthesis (TEP), abdomen/groin hernia) or diseases (i.e. epilepsy, cardiac arrhythmia) that prevent WB-EMS intervention
* medication and/or diseases affecting our primary endpoints.

Min Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Appendicular skeletal muscle mass | baseline - 6 months follow-up
  changes of appendicular skeletal muscle mass from baseline to 6 month follow-up
Muscle density of the medial thigh | baseline - 6 months follow-up
  changes of muscle density (thigh) from baseline to 6 month follow-up
Intramuscular fat content | baseline - 6 months follow-up
  changes of Intramuscular fat content (thigh) from baseline to 6 month follow-up

SECONDARY OUTCOMES:
Muscle cross sectional area (CSA) | baseline - 6 months follow-up
  changes of muscle CSA (thigh) from baseline to 6 month follow-up
Isokinetic leg strength | baseline - 6 months follow-up
  changes of isokinetic leg strength from baseline to 6 month follow-up
Short Physical Performance Battery (SPPB) | baseline - 6 months follow-up
  SPPB according to Guralnik et al. (J Gerontol Med Sci1994; 49(2):M85-M94)
Hand grip of the dominant hand | baseline - 6 months follow-up
  Maximum isometric strength of the dominant hand (dynamometer)
muscular power of the legs | baseline - 6 months follow-up
  Muscular power of the legs (jumping test), by Leonardo (Novotec, Germany)

OTHER OUTCOMES:
Balance according to SPPB | baseline - 6 months follow-up
  Balance according to SPPB (see above), Soehnle balance platform device (Soehnle Germany)
Quality of life | baseline - 6 months follow-up
  Quality of Life: EUROQuOI questionnaire
Trial Making Tests A and B | baseline - 6 months follow-up
  TMT-L: Trail Making Test - Langensteinbacher version.

CONTACTS AND LOCATIONS:
Overall Officials: Cornel Sieber, MD, Study Chair — Institute of Biomedicine of Age, University of Erlangen-Nuremberg; Cornelius Bollheimer, MD, Study Chair — Institute of Biomedicine of Age, University of Erlangen-Nuremberg; Klaus Engelke, PhD, Study Director — Institute of Medical Physics, University of Erlangen-Nuremberg; Wolfgang Kemmler, PHD, Principal Investigator — Institute of Medical Physics, University of Erlangen-Nuremberg; Ellen Freiberger, PhD, Principal Investigator — Institute of Biomedicine of Age, University of Erlangen-Nuremberg

REFERENCES:
- [Background] Kemmler W, Bebenek M, Engelke K, von Stengel S. Impact of whole-body electromyostimulation on body composition in elderly women at risk for sarcopenia: the Training and ElectroStimulation Trial (TEST-III). Age (Dordr). 2014 Feb;36(1):395-406. doi: 10.1007/s11357-013-9575-2. Epub 2013 Aug 16. PMID 23949160
- [Background] Kemmler W, von Stengel S. Whole-body electromyostimulation as a means to impact muscle mass and abdominal body fat in lean, sedentary, older female adults: subanalysis of the TEST-III trial. Clin Interv Aging. 2013;8:1353-64. doi: 10.2147/CIA.S52337. Epub 2013 Oct 7. PMID 24130433
- [Derived] Kemmler W, Teschler M, Weissenfels A, Bebenek M, von Stengel S, Kohl M, Freiberger E, Goisser S, Jakob F, Sieber C, Engelke K. Whole-body electromyostimulation to fight sarcopenic obesity in community-dwelling older women at risk. Resultsof the randomized controlled FORMOsA-sarcopenic obesity study. Osteoporos Int. 2016 Nov;27(11):3261-3270. doi: 10.1007/s00198-016-3662-z. Epub 2016 Jun 12. PMID 27289534